CLINICAL TRIAL: NCT02427295
Title: Long-term (up to 3 Years) Clinical and Hormonal Outcomes in Acromegalic Patients With Treated Surgery With or Without Long Acting Somatostatin Analogues: Open-labeled, Prospective, Parallel Group Study
Brief Title: Hormonal Outcomes in Acromegalic Patients With Treated Surgery With or Without Long Acting Somatostatin Analogues
Acronym: acromegaly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis Korea Ltd. (Industry)
Responsible Party: Principal Investigator, min seon kim, principal investigator, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMS995BKR08T
Record Dates: First submitted 2015-02-04; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 2: Surgery + Medical treatment (Experimental): MRI : residual tumor 6 months post-op : IGF-1 >600 ng/ml
  medical treatment : Sandostatin (Octreotide Acetate)
  Interventions: Drug: Sandostatin (Octreotide Acetate)
- Group 3 : Rescue group (No Intervention): If IGF-1 levels fails to normalize till post-op 18 months post-op, medical treatment will be added.)
- Gruop1 : Surgery only group (No Intervention): MRI : without residual tumor 6months post-operation
  and IGF-1 <600ng/ml

INTERVENTIONS:
Drug: Sandostatin (Octreotide Acetate) — For the patients outlined above (refer to 2), subjects who are not able to be treated by surgery alone:
  * Dose: Sandostatin LAR® 20mg per 4 weeks for 3 months -> If serum IFG-1 levels fails to normalize, the dose of LAR will be increased to 30 mg.
  * Frequency: every 4 weeks.
  * Route of administration: IM injection.
  Other Names: Sandostatin LAR
  Arms: Group 2: Surgery + Medical treatment

SUMMARY:
Long-term (up to 3 years) clinical and hormonal outcomes in acromegalic patients with treated surgery with or without long acting somatostatin analogues.

DETAILED DESCRIPTION:
Patients who are diagnosed with acromegaly with a GH-secreting pituitary adenoma receiving TSA at the Asan Medical Center (Seoul, Korea) from Aug 2013 to Aug 2015 will be recruited.

The eligible patient population will consist of 30 adult, male and female patient with Age 18 or older.

* Number of patients by treatment group: Surgical treatment only = 15, Surgery with medical treatment = 15
* Number of Centers: 1 (single center)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Patients diagnosed with acromegaly with GH-secreting pituitary adenoma on sellar MRI, meeting the biochemical criteria outlined above (refer to 1. Diagnosis of acromegaly) and with typical acromegalic features.
3. No prior use of somatostatin analogues.
4. Adequate hepatic and renal function
5. Provision of a signed written informed consent

Exclusion Criteria:

1. Severe co-morbid illness such as untreatable other malignancy and/or active infections.
2. Pregnant or lactating women
3. Hypersensitivity to Sandostatin or any component of the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieved normalization of fasting serum IGF-1 (age and sex matched) | Change from within 3days post-operative in fasting serum IGF-1at 36 months post-operative
The time taken to IGF-1 normalization in each group. | Change from within 3days post-operative in IGF-1 normalization at 36 months post-operative months post-operative

SECONDARY OUTCOMES:
GH suppressive responses (a nadir GH < 0.4 ng/ml) to oral glucose | Change from Pre-operative in GH suppressive responses (a nadir GH < 0.4 ng/ml) at 36 months post-operative
Clinical symptom and sign with AcroQoL questionnaire | Change from Pre-operative in Clinical symptom and sign with AcroQoL questionnaire at 36 months post-operative
Sleep quality and disturbance with written questionnaire | Change from Pre-operative in Sleep quality and disturbance with written questionnaire at 24 months post-operative
fasting glucose , postprandial glucose | Change from pre-operative in fasting glucose , postprandial glucose at 36 months post-operative.
insulin | Change from pre-operative in insulin at 36 months post-operative.
HbA1c | change from pre-operative in HbA1c at 36 months post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: minseon Kim, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea